CLINICAL TRIAL: NCT04526015
Title: The Analgesic Effect of Iliohypogastric and Ilioinguinal Nerve Block for Acute and Chronic Pain Relief After Cesarean Section Delivery.Randomized Controlled Study Post
Brief Title: Iliohypogastric and Ilioinguinal Nerve Block for Acute and Chronic Pain Relief After Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain relief for c.s
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Iliohypogastric and Ilioinguinal Nerve Block for Acute and Chronic Pain in Cesarean Section

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilioinguinal iliohypogastric Block (Experimental): Each patient will receive spinal anesthesia plus bilateral ultrasound-guided IL/IH nerve block. The abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualized between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side
  Interventions: Procedure: Iliohypogastric and ilioinguinal nerve block
- Controlled Group (Other): Each patient will receive spinal anesthesia alone with no block.
  Interventions: Procedure: Controlled Group

INTERVENTIONS:
Procedure: Iliohypogastric and ilioinguinal nerve block — Each patient will receive spinal anesthesia plus bilateral ultrasound-guided IL/IH nerve block. The abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualized between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side
  Arms: Ilioinguinal iliohypogastric Block
Procedure: Controlled Group — Each patient will receive spinal anesthesia alone with no block.
  Arms: Controlled Group

SUMMARY:
The increase in CS in recent years makes even a small prevalence of persistent pain after CS a significant burden, both financially and in terms of quality of life, for a large number of otherwise healthy young women. Persistent pain after CS has been shown to be associated with postpartum depression, interferes with daily activities, and causes sleep disturbances, all of which negatively and directly impact the mother. As a result, the care of the baby by the mother is affected negatively.

To adequately control postoperative pain, healthcare providers use a one-size-fits-all multimodal analgesic approach and sensible opioid prescription with monitoring to prevent addiction. The challenge is in tailoring this approach to the outliers who may be opioid tolerant or opioid-sensitive. However, the severity and duration of postoperative pain and its management may be predictive of developing persistent pain at two to 12 months or later.

Previous studies revealed different outcomes regarding the analgesic efficacy of II-IH nerve block for post caesarean pain, inguinal repair and surgery involving the female genital tract. Moreover, exploring the efficacy of II-IH nerve block could help to tackle sever postoperative pain after cesarean delivery particularly in settings where there is shortage of epidural kit supply and availability of strong opioids for pain management. We aimed to assess the analgesic efficacy of bilateral ilioinguinal and iliohypogastric nerve block for planned caesareans delivery under spinal anaesthesia and evaluate the incidence of persistent pain with transition from acute to chronic pain.

DETAILED DESCRIPTION:
All patients will be assessed preoperatively by history taking, physical examination, and laboratory evaluation. On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure and pulse oximetry will be applied.

The patients will be positioned in sitting position to give the spinal anesthesia at L3-L4/L2-L3 intervertebral level in the midline approach. After local infiltration of skin and subcutaneous tissue with 2% lignocaine, 25 G B-braun spinal needle will be used to administer subarachnoid block (SAB) with 2.5 ml of hyperbaric bupivacaine (5%) and 20 µg of fentanyl after confirmation of free flow of cerebrospinal fluid (CSF) at the hub of the needle. Patients will be coloaded with 10-12 ml/kg (over the period of 15 min) of Ringer's Lactate (RL) solution at the time of SAB. Thereafter, patients will be placed in supine position with wedge under the right hip.

64 Patients were randomly allocated into two equal groups (each 32 patients):

* Group B (IL/IH group): Each patient will receive spinal anesthesia plus bilateral ultrasound-guided IL/IH nerve block. The abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualized between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side
* Group C (Controlled group): Each patient will receive spinal anesthesia alone with no block.

Postoperative Analgesia Protocol

All patients will be given a standardized patient controlled intravenous analgesia (PCIA) regimen. The disposable PCIA device (Coopdech Syrinjector PCA set; Daiken Medical) contained 30 mg morphine in 45 ml saline. Patients will be instructed on how to use the PCIA device, which was set with a bolus of 2 mg morphine and a minimum interval of 30 min. If the analgesic effect was not satisfactory, complementary use of intravenous morphine will be applied.

Assessment of Acute Postoperative Pain

At 24 hours after surgery, pain intensity will be recorded on a 10-point verbal pain rating scale ranging from 0 to 10 (VPRS; 0 = no pain to 10 = worst pain imaginable), at rest (VPRS-R) and while moving into the sitting position (VPRS-S). Pain will be considered none, mild, moderate, or severe if scored 0, 1 to 3, 4 to 6, or 7 to 10, respectively.

Assessment of Persistent Postoperative Pain (3 and 6 Months) The Short-Form McGill Pain Questionnaire-Revised (SFMPQ- 2) was designed specifically and validated to assess both neuropathic and non-neuropathic aspects of chronic pain.

Women will report their average and worst pain the week prior to and at the time of the telephone interview using a previously developed scripted telephone interview. Persistent pain will be defined as new onset of pain related to the CS, located around the scar or in the abdomen, and still present at 8 weeks. Chronic pain will be defined if same symptoms were still present at 3 and 6 months.

Measurements The following parameters will be recorded by an anesthesia resident not included in the study and blinded to its groups: -

* Demographic data (Age in month, body mass index, and ASA class)
* Total consumption of analgesia (mg/kg) in first day postoperatively. (Primary outcome)
* The time to the first rescue analgesic request. (Secondary outcome) The postoperative pain score (NRS pain score). Assessment of the presence and intensity of pain was done immediately after transfer to the ward (0 h) and at 4 h, 6 h , 12 h and 24 h after surgery both at rest and with movement (turning from side to side) by using verbally administered Numerical rating scale pain assessment tools.
* The incidence of perioperative complications including bradycardia, hypotension, nausea and vomiting, localized hematoma, infection, or pruritis.
* Incidence of chronic pain at 3 & 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female.less than 40 years .
* ASA l,ll full term scheduled for elective cesarean section

Exclusion Criteria:

* patient refusal
* Emergency section
* More than I prior section
* Current pain disorder
* Allergy to local anesthetic
* Coagulopathy
* Major cardiac,renal, hepatic disorder

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The total dose of morphine used Patients rescue analgesia within first 24h postoperative | up to 24 hours postoperative
  The total dose of morphine used postoperatively/patient (rescue analgesia) within first 24 h postoperative

SECONDARY OUTCOMES:
Incidence of chronic pain at 3 & 6 months. | up to 6 months
  Incidence of chronic pain at 3 & 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ELgharbiaa, Egypt